CLINICAL TRIAL: NCT06469281
Title: A Phase 1a/1b Study of 27T51, an Anti-MUC16 CAR T Cell Drug Product Administered Alone or in Combination for Participants With Recurrent or Refractory Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Brief Title: A Study to Learn if 27T51, a Mucin-16 (MUC16) Protein Targeting Immune Cell Therapy, Administered Alone or in Combination is Safe and How Well it Works for Adult Participants With Recurrent or Treatment Resistant Ovarian Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 27T51-01
Record Dates: First submitted 2024-06-06; First posted 2024-06-21 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Epithelial Ovarian Cancer; Primary Peritoneal Carcinoma; Fallopian Tube Cancer
Keywords: Ovarian Cancer; CAR T; Peritoneal; Fallopian Tube; MUC16; Immunotherapy
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — cemiplimab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation (Experimental): 27T51 monotherapy
  Interventions: Other: 27T51
- Dose Expansion - Arm A (Experimental): 27T51 monotherapy
  Interventions: Other: 27T51
- Dose Expansion - Arm B (Experimental): 27T51+Cemiplimab
  Interventions: Other: 27T51; Drug: Cemiplimab
- Dose Expansion - Arm C (Experimental): 27T51+Cemiplimab+Bevacizumab
  Interventions: Other: 27T51; Drug: Cemiplimab; Drug: Bevacizumab

INTERVENTIONS:
Other: 27T51 — Intravenous (IV) infusion
Drug: Cemiplimab — IV infusion
  Other Names: Libtayo; REGN2810
  Arms: Dose Expansion - Arm B; Dose Expansion - Arm C
Drug: Bevacizumab — IV Infusion
  Other Names: Avastin; Mvasi; Vegzelma; Zirabe
  Arms: Dose Expansion - Arm C

SUMMARY:
This study is researching an experimental CAR T cell therapy called 27T51, referred to as study drug. The study drug is a MUC16 targeting immune cell therapy focused on adult female participants with recurrent or difficult to treat epithelial ovarian, primary peritoneal or fallopian tube cancer.

This study has two (2) major parts:

Phase 1a Dose Escalation and Phase 1b Dose Expansion. The aim of the dose escalation part will be to test the safety of 27T51 in a small number of participants to find the highest dose given to humans without unacceptable side effects. The aim of the dose expansion part will be to test 27T51 at the established dose level(s) from the dose escalation part and may include other medications given in combination with 27T51.

Information collected from this study will help researchers understand more fully whether this immune cell therapy, also known as CAR T cell therapy, can be safely used to treat solid tumors such as ovarian cancer.

DETAILED DESCRIPTION:
Former Sponsor 2seventy bio

ELIGIBILITY:
Key Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
2. Histological diagnosis of epithelial ovarian, primary peritoneal, or fallopian tube cancer according to World of Health Organization (WHO) 2020 classification
3. Recurrent or refractory epithelial ovarian, primary peritoneal, or fallopian tube cancer, as described in the protocol
4. Serum cancer antigen (CA) 125 ≥ 2 × upper limit of normal (ULN) as assessed at the local lab by a 510(k) cleared test at screening
5. Participants must have at least 1 measurable tumor lesion as defined by the response evaluation criteria in solid tumors (RECIST) 1.1.
6. Expected survival ≥ 3 months

Key Exclusion Criteria:

1. Inadequate cardiovascular, renal and hepatic function, as described in the protocol
2. Absolute lymphocyte count (ALC) < 100 cells/μL at time of leukapheresis
3. History of Grade ≥ 2 hemorrhage within 30 days, or inadequate coagulation parameters, as described in the protocol
4. Known history or presence of clinically relevant central nervous system (CNS) pathology, as described in the protocol
5. Ongoing or recent (within 2 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk for immune related adverse events (AEs)
6. Treatment with any cellular or gene therapy

Note: Other protocol-defined Inclusion/Exclusion criteria apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2030-05-27 (Estimated); Study Completion 2030-05-27 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) | Up to 18 months
  Part 1a
Incidence of adverse events of special interest (AESIs) | Up to 18 months
  Part 1a
Incidence of adverse events of dose limiting toxicities (DLTs) | Up to 18 months
  Part 1a
Manufacturing feasibility of 27T51 | Up to 3 years
  Phase 1a/1b Determination of the feasibility of manufacturing 27T51 is measured by the percent of leukapheresis products collected that are able to be manufactured and released for infusion.
Overall response rate (ORR) as assessed by the investigator | Up to 48 months
  Phase 1b

SECONDARY OUTCOMES:
ORR as assessed by the investigator | Up to 48 months
  Phase 1a
Duration of response (DoR) | Up to 48 months
  Phase 1a/1b
Disease control rate (DCR) | Up to 48 months
  Phase 1a/1b
Incidence of TEAEs | Up to 48 months
  Phase 1b
Incidence of AESIs | Up to 48 months
  Phase 1b
Incidence of DLTs | Up to 48 months
  Phase 1b - Arms B and C

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (5):
- United States (5):
  - Massachusetts General Hospital, Boston, Massachusetts
  - John Theurer Cancer Center Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - LDS Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/